CLINICAL TRIAL: NCT05030753
Title: iSIPsmarter: An RCT to Evaluate the Efficacy, Reach, and Engagement of a Technology-based Behavioral and Health Literacy Intervention to Reduce Sugary Beverages Among Rural Appalachian Adults
Brief Title: iSIPsmarter: An RCT Evaluating the Efficacy of a Technology-Based Intervention to Reduce Sugary Drinks in Rural Appalachia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: University of North Carolina (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Jamie Zoellner, PhD RD, Director, Community Based Health Equity Program, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: University of Virginia; R01MD015033 (NIH)
Record Dates: First submitted 2021-08-13; First posted 2021-09-01 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-09

CONDITIONS: Diet Habit; Sugar-Sweetened Beverages
Keywords: sugar-sweetened beverages; weight; rural; health disparities; self-monitoring; internet intervention; e/m health; test messaging
MeSH Terms: conditions — Feeding Behavior; Body Weight | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iSIPsmarter (Experimental): iSIPsmarter is a technology-based behavioral and health literacy intervention. It is comprised of six Internet-delivered Cores, an integrated short message service (SMS) strategy to engage users in tracking SSB behaviors, and the incorporation of a cellular enabled scale for in-home weight tracking. Participants will be prompted (via email or text) to self-monitor their sugar-sweetened beverage intake. iSIPsmarter is a highly interactive, structured, and self-guided program that uses strategies previously proven to promote behavior change. iSIPsmarter also incorporates a stepped care approach to re-engage users who struggle to complete components.
  Interventions: Behavioral: iSIPsmarter
- Patient Education (PE) (Active Comparator): he PE website will include scientifically accurate information that is typical of nutrition education websites and will include information about SSB recommendations, types of SSB and portion size, SSB-related health risks, energy balance information, identifying personal motivators and barriers to reducing SSB intake, interpreting SSB nutrition labels, and recognizing media influences and misclaims in SSB advertisements, as well as printable forms to track SSB and weight. Unlike iSIPsmarter, the content will not be tailored and will be presented all at once.
  Interventions: Behavioral: Patient Education (PE)

INTERVENTIONS:
Behavioral: iSIPsmarter — iSIPsmarter is a technology-based behavioral and health literacy intervention. It is comprised of six Internet-delivered Cores, an integrated short message service (SMS) strategy to engage users in tracking SSB behaviors, and the incorporation of a cellular enabled scale for in-home weight tracking. Participants will be prompted (via email or text) to self-monitor their sugar-sweetened beverage intake. iSIPsmarter is a highly interactive, structured, and self-guided program that uses strategies previously proven to promote behavior change. iSIPsmarter also incorporates a stepped care approach to re-engage users who struggle to complete components.
  Arms: iSIPsmarter
Behavioral: Patient Education (PE) — he PE website will include scientifically accurate information that is typical of nutrition education websites and will include information about SSB recommendations, types of SSB and portion size, SSB-related health risks, energy balance information, identifying personal motivators and barriers to reducing SSB intake, interpreting SSB nutrition labels, and recognizing media influences and misclaims in SSB advertisements, as well as printable forms to track SSB and weight. Unlike iSIPsmarter, the content will not be tailored and will be presented all at once.
  Arms: Patient Education (PE)

SUMMARY:
The proposed randomized controlled trial (RCT) is guided by the RE-AIM (i.e. reach, efficacy, adoption, implementation, maintenance) framework and targets 244 adults from rural Appalachia. The overall goal is to examine the efficacy of iSIPsmarter in a 2 group [iSIPsmarter vs. static Patient Education (PE) website] by 4 assessment (Pre, 3-, 6- and 18-month follow-up) design. It is hypothesized that iSIPsmarter will be more efficacious at reducing SSB consumption than a PE website at post assessment.

DETAILED DESCRIPTION:
Sugar-sweetened beverages (SSB, e.g., soda/pop, sweet tea, sports and energy drinks, fruit drinks) are the largest single food source of calories in the United States (US) diet and contributes approximately 7% of total daily energy intake for US adults. Among Appalachian adults, SSB intake is disproportionately high, averaging about 14% of total daily energy intake. There are strong and consistent data documenting relationships among high SSB consumption and numerous health issues such obesity, diabetes, some obesity-related cancers, coronary heart disease, hypertension, and dental decay. Further compounding the SSB problem, the Appalachian region lacks access to providers, medical services, and evidence-based behavioral prevention programs. There is also limited data on technology-based behavioral interventions in Appalachia. However, given recent progress in shrinking the digital divide, the timing is optimal to evaluate technology-based behavioral interventions in this region. The current proposal is designed to target this major SSB dietary risk factor and public health challenge, as well as address notable gaps in the rural e/m-Health literature. Importantly, this proposal builds on our team's e/m-Health intervention expertise and decade of SSB behavioral intervention research in rural Appalachia. iSIPsmarter is a technology-based behavioral and health literacy intervention targeting SSB reduction and weight reduction/maintenance. It is comprised of six core Internet-delivered modules, an integrated short message service (SMS) strategy to engage users in tracking SSB behaviors, and a cellular enabled scale for in-home weight tracking. iSIPsmarter is a highly interactive, structured, and self-guided program that uses strategies previously proven to promote behavior change. iSIPsmarter also incorporates a stepped care approach to engage users who struggle to complete components of the intervention. The proposed RCT is guided by the RE-AIM framework and targets 244 adults from rural Appalachia. The overall goal is to examine the efficacy of iSIPsmarter in a 2 group [iSIPsmarter vs. static Patient Education (PE) website] by 4 assessment (Pre, 3-, 6- and 18-month follow-up) design. It is hypothesized that iSIPsmarter will be more efficacious at reducing SSB consumption than a PE website at post assessment. Changes in secondary outcomes (e.g. overall dietary quality, weight, quality of life) and maintenance of outcomes at 6- and 18-months post intervention will also be evaluated. Additional secondary aims include to examine reach and representativeness, patterns of user engagement, and cost. Two tertiary aims include exploratory mediation analyses and a systems-level, participatory process to understand context for future organizational-level adoption of iSIPsmarter, and specifically to explore factors that would promote or inhibit a sustainable SSB screening and referral process. The long-term goal of this line of this research is to sustain an effective, scalable, and high reach behavioral intervention to improve SSB behaviors and weight and to reduce SSB-related health inequities and chronic conditions in rural Appalachia and beyond.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults, > or equal to 18 years of age, consume >200 kcals of SSB/day, ability and willingness to access an internet-enabled device at least one time per week and receive SMS-based reminder prompts.

Exclusion Criteria:

* non-English speaking adults, <18 years of age, consume <200 kcals of SSB/day, inability and willingness to access an internet-enabled device at least one time per week and receive SMS-based reminder prompts. Also, only one person per household is eligible to participate in the trial.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie M Zoellner, PhD, Principal Investigator — University of Virginia; Lee Ritterband, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zoellner JM, You W, Porter K, Reid AL, Brock DP, Markwalter T, Frederick C, Tate DF, Ritterband L. A digital behavioral intervention to reduce sugar-sweetened beverage consumption: a randomized, controlled trial. Am J Clin Nutr. 2025 Aug;122(2):544-555. doi: 10.1016/j.ajcnut.2025.06.010. Epub 2025 Jun 11. PMID 40513952
- [Derived] Zoellner JM, Porter KJ, You W, Reid AL, Frederick C, Hilgart M, Brock DP, Tate DF, Ritterband LM. Study protocol for iSIPsmarter: A randomized-controlled trial to evaluate the efficacy, reach, and engagement of a technology-based behavioral intervention to reduce sugary beverages among rural Appalachian adults. Contemp Clin Trials. 2021 Nov;110:106566. doi: 10.1016/j.cct.2021.106566. Epub 2021 Sep 4. PMID 34492306

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | iSIPsmarter | Patient Education (PE)
Started | 127 | 122
Completed | 127 | 122
Not Completed | 0 | 0
Period: 9-week
Arm/Group | iSIPsmarter | Patient Education (PE)
Started | 127 | 122
Completed | 114 | 114
Not Completed | 13 | 8
Not completed — Lost to Follow-up | 10 | 7
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Excluded from analysis due to missing covariates | 2 | 1
Period: 6-month post intervention
Arm/Group | iSIPsmarter | Patient Education (PE)
Started | 114 | 114
Completed | 105 | 110
Not Completed | 9 | 4
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by Subject | 4 | 0
Period: 18-month post intervention
Arm/Group | iSIPsmarter | Patient Education (PE)
Started | 105 | 110
Completed | 102 | 109
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | iSIPsmarter | Patient Education (PE) | Total
Number analyzed (Participants) | 127 | 122 | 249
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 125 | 116 | 241
  >=65 years | 2 | 6 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (13.2) | 41.2 (13.2) | 41.6 (12.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 24 | 17 | 41
  Female | 103 | 104 | 207
  Other | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 121 | 118 | 239
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 4 | 13
  White | 113 | 108 | 221
  More than one race | 2 | 6 | 8
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 127 | 122 | 249
Annual Household Income [Count of Participants; unit: Participants]
  <= $14,999 | 9 | 8 | 17
  $15,000-$34,999 | 27 | 22 | 49
  $35,000-$54,999 | 26 | 36 | 62
  >= $55,000 | 63 | 56 | 119
  Unknown or unreported | 2 | 0 | 2
Education Level, categorical [Count of Participants; unit: Participants]
  <= High school graduate | 14 | 9 | 23
  Some college or greater | 113 | 113 | 226
Perceived Health Literacy, continuous [Mean (Standard Deviation); unit: units on a scale] — 3 single-item subjective rating of Health literacy reported on a 5-point Likert scale and summed to create a total score ranging from 0 to 12. Questions include confidence in completing medical forms on their own, needing help with written medical instructions and other materials, and overall reading abilty. Higher scores indicate higher levels of health literacy.
  units on a scale | 11.6 (1.00) | 11.5 (0.99) | 11.5 (0.99)
Rurality Status, categorical [Count of Participants; unit: Participants] — Determined by county level Rural Urban Continuum Codes (RUCC). Ranges from 1-9 with higher scores indicating greater rurality. For the study, the RUCC codes were broken down into three categories: 1-2=large to medium metro areas, 3=small metro areas with overlapping rural and urban characteristics, and 4-9=non metro or rural areas.
  Participants
    RUCC 1-2 | 16 | 20 | 36
    RUCC 3 | 57 | 54 | 111
    RUCC 4-9 | 54 | 48 | 102
Weight, continuous [Mean (Standard Deviation); unit: kilograms] — Weight obtained during enrollment via a cellular enabled BodyTrace scale. Weight was retrieved by researchers via the BodyTrace online interface. Population: 10 participants were excluded from analysis due to missing weight data (n=1), defective scales (n=4), pregnancy (n=2), bariatric surgery (n=1), and exceeding the scales maximum weight (n=2)
  kilograms
    number analyzed (Participants) | 122 | 117 | 239
    (all) | 94.2 (26.8) | 90.6 (23.6) | 92.4 (25.4)
BMI, continuous [Mean (Standard Deviation); unit: kg/m^2] — Population: 10 participants were excluded from analysis due to missing weight data (n=1), defective scales (n=4), pregnancy (n=2), bariatric surgery (n=1), and exceeding the scales maximum weight (n=2)
  kg/m^2
    number analyzed (Participants) | 122 | 117 | 239
    (all) | 33.8 (9.0) | 32.5 (8.0) | 33.2 (8.7)
BMI, categorical [Count of Participants; unit: Participants] — BMI categorized according to the CDC guidelines: <=18.4=underweight, 18.5-24.9=normal weight, 25-29.9=overweight, 30-34.9=obesity I, 35-39.9=obestity II, >=40=obesity III. Population: 10 participants were excluded from analysis due to missing weight data (n=1), defective scales (n=4), pregnancy (n=2), bariatric surgery (n=1), and exceeding the scales maximum weight (n=2)
  Participants
    number analyzed (Participants) | 122 | 117 | 239
    Underweight | 0 | 1 | 1
    Overweight | 17 | 22 | 39
    Normal | 30 | 28 | 58
    Obesity Class 1 | 28 | 27 | 55
    Obesity Class 2 | 19 | 19 | 38
    Obesity Class 3 | 28 | 20 | 48
Sugar-sweetened beverage fluid milliliters/day [Mean (Standard Deviation); unit: fluid milliliters/day] — The primary sugar-sweetened beverage (SSB) outcome was assessed with the BEVQ-15, which queries intake over the past 30 days. Using standardized and validated scoring procedures, totals for the five SSB-related beverages (i.e., regular soft drinks, sweetened juice beverage/drink, sweetened tea, coffee with sugar, energy/sports drinks) were determined by multiplying reported intake frequency by portion size, and then summing the five categories to obtain total daily intake of all SSB.
  fluid milliliters/day | 1313.1 (760.0) | 1144.5 (603.3) | 1230.2 (692.0)
Sugary-sweetened beverage kilocalories/day [Mean (Standard Deviation); unit: kilocalories/day] — The primary sugar-sweetened beverage (SSB) outcome was assessed with the BEVQ-15, which queries past 30 day intake. Using standardized and validated scoring procedures, totals for the five SSB-related beverages (i.e., regular soft drinks, sweetened juice beverage/drink, sweetened tea, coffee with sugar, energy/sports drinks) were determined by multiplying reported intake frequency by portion size, and then summing the five categories to obtain total daily intake of all SSB. Standardized kilocaloried information for the drink categories were used to determine estimates of daily SSB kcal.
  kilocalories/day | 514.4 (317.5) | 446.2 (249.7) | 481.0 (287.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Sugar-sweetened Beverage Fluid Milliters/Day at 9-weeks
Description: The primary sugar sweetened beverage (SSB) outcome was assessed with the BEVQ-15, which queries intake over the past 30 days. Using standardized and validated scoring procedures, totals for the five SSB-related beverages (i.e., regular soft drinks, sweetened juice beverage/drink, sweetened tea, coffee with sugar, energy/sports drinks) were determined by multiplying reported intake frequency by portion size, and then summing the five categories to obtain total fluid milliters/day intake of all SSB.
Time Frame: Baseline, 9-weeks (immediate-post follow-up)
Population: Participants who completed Baseline and 9-week Bev-Q survey, were not previously lost to follow-up or withdrawn from the study, and had complete data for covariates used in the analysis (age, sex, race, income, educational level, and health literacy).
Measure: Least Squares Mean (95% Confidence Interval); unit: fluid milliters/day
Arm/Group | iSIPsmarter | Patient Education (PE)
Number analyzed (Participants) | 114 | 114
fluid milliters/day | -897.0 [-1044.2 to -749.4] | -291.0 [-493.9 to -88.1]

2. Secondary Outcome: Change From Baseline Sugar-sweetened Beverage Fluid Milliters/Day at 6-months Post Intervention
Description: as for outcome 1
Time Frame: Baseline, 6-months (post-intervention follow-up)
Population: Participants who completed the Bev-Q at 6-months, were not previously lost to follow-up or withdrawn from the study, and had complete data for covariates used in the analysis (age, sex, race, income, educational level, and health literacy).
Measure: Least Squares Mean (95% Confidence Interval); unit: fluid milliters/day
Arm/Group | iSIPsmarter | Patient Education (PE)
Number analyzed (Participants) | 105 | 110
fluid milliters/day | -858.2 [-1008.2 to -708.3] | -279.5 [-490.3 to -68.6]

3. Secondary Outcome: Change From Baseline Sugar-sweetened Beverage Fluid Milliters/Day at 18-months Post Intervention
Description: The primary sugar sweetened beverage (SSB) outcome was assessed with the BEVQ-15, which queries intake over the past 30 days. Using standardized and validated scoring procedures, totals for the five SSB-related beverages (i.e., regular soft drinks, sweetened juice beverage/drink, sweetened tea, coffee with sugar, energy/sports drinks) were determined by multiplying reported intake frequency by portion size, and then summing the five categories to obtain total fluid milliters/day of all SSB.
Time Frame: Baseline, 18-months (post itnervention follow-up)
Population: Participants who completed the Bev-Q at 18-months, were not previously lost to follow-up or withdrawn from the study, and had complete data for covariates used in the analysis (age, sex, race, income, educational level, and health literacy).
Measure: Least Squares Mean (95% Confidence Interval); unit: fluid milliters/day
Arm/Group | iSIPsmarter | Patient Education (PE)
Number analyzed (Participants) | 102 | 109
fluid milliters/day | -893.1 [-1044.5 to -737.0] | -618.7 [-762.1 to -475.2]

4. Secondary Outcome: Percent Weight Change From Baseline Weight at 9-weeks
Description: Using weight data collected from a cellular enabled in-home ©BodyTrace digital scale and calculating percent weight change between Baseline and 9-weeks (immediate post follow-up).
Time Frame: Baseline, 9-weeks (immediate-post follow-up)
Population: Participants who weighed themselves on the BodyTrace scale, did not have an excluded weight (e.g., pregnancy, defective scale, bariatric surgery, weight exceed scale limit), were not lost to follow-up or withdrawn from the study, and had complete data for covariates used in the analysis (age, sex, race, income, educational level, and health literacy).
Measure: Least Squares Mean (95% Confidence Interval); unit: percent weight change
Arm/Group | iSIPsmarter | Patient Education (PE)
Number analyzed (Participants) | 107 | 108
percent weight change | -1.13 [-1.84 to -0.42] | -0.05 [-0.36 to 0.26]

5. Secondary Outcome: Percent Weight Change From Baseline Weight at 6-months
Description: Using weight data collected from a cellular enabled in-home ©BodyTrace digital scale and calculating percent weight change between Baseline and 6-months (post intervention follow-up).
Time Frame: Baseline, 6-months (post-intervention follow-up)
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percent weight change
Arm/Group | iSIPsmarter | Patient Education (PE)
Number analyzed (Participants) | 100 | 101
percent weight change | -1.95 [-3.34 to -0.55] | -0.55 [-1.74 to 0.64]

6. Secondary Outcome: Percent Weight Change From Baseline Weight at 18-months
Description: as for outcome 5
Time Frame: Baseline, 18-months (post-intervention follow-up)
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percent weight change
Arm/Group | iSIPsmarter | Patient Education (PE)
Number analyzed (Participants) | 88 | 91
percent weight change | -2.97 [-4.48 to -1.45] | -0.000003 [-0.00002 to 0.00000833]

7. Secondary Outcome: Change From Baseline Overall Quality of Life at 9-weeks
Description: Using the Center's for Disease (CDC) Healthy Days Core Module to measure total days in the past month that were either physically or mentally unhealth. Range is from 0-30. Lower scores indicate greater quality of life.
Time Frame: Baseline, 9-weeks (immediate post-folllow-up)
Population: Participants who completed the Healthy Days scale, were not lost to follow-up or withdrawn from the study, and had complete data for covariates used in the analysis (age, sex, race, income, educational level, and health literacy).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | iSIPsmarter | Patient Education (PE)
Number analyzed (Participants) | 113 | 113
score on a scale | -0.61 [-3.32 to 2.11] | -1.28 [-3.90 to 1.34]

8. Secondary Outcome: Change From Baseline Overall Quality of Life at 6-months
Description: as for outcome 7
Time Frame: Baseline, 6-months (post intervention follow-up)
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | iSIPsmarter | Patient Education (PE)
Number analyzed (Participants) | 104 | 109
score on a scale | -5.08 [-7.50 to -2.66] | -5.31 [-7.80 to -2.83]

9. Secondary Outcome: Change From Baseline Overall Quality of Life at 18-months
Description: as for outcome 7
Time Frame: Baseline, 18-months (post intervention follow-up)
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | iSIPsmarter | Patient Education (PE)
Number analyzed (Participants) | 101 | 107
score on a scale | -0.71 [-3.62 to 2.21] | -1.92 [-4.79 to 0.95]

10. Secondary Outcome: Change From Baseline Dietary Quality as Measured by the Healthy Eating Index (HEI) Score at 9-weeks
Description: 2 unannounced recalls (one weekend and one weekday) using state-of-the-art Nutrition Data System for Research (NDSR) software and multiple pass methods. HEI indicators will be extracted from the NDSR system and examined for changes in the total HEI score, on a 100-point continuous scale (higher scores reflective higher diet quality).
Time Frame: Baseline, 9-weeks (immediate-post follow-up)
Population: Participants who completed dietary recalls at all time points (Baseline, 9-weeks, 6-months, and 18 months).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | iSIPsmarter | Patient Education (PE)
Number analyzed (Participants) | 100 | 108
score on scale | 1.70 [-1.13 to 4.52] | 2.82 [-0.06 to 5.70]

11. Secondary Outcome: Change From Baseline Dietary Quality as Measured by the Healthy Eating Index (HEI) Score at 6-months
Description: as for outcome 10
Time Frame: Baseline, 6-months (post intervention follow-up)
Population: Participants who completed dietary recalls at all time points (Baseline, 9-weeks, 6-months, and 18 months).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | iSIPsmarter | Patient Education (PE)
Number analyzed (Participants) | 100 | 108
score on a scale | 3.33 [0.56 to 6.11] | 1.65 [-1.00 to 4.30]

12. Secondary Outcome: Change From Baseline Dietary Quality as Measured the Healthy Eating Index (HEI) Score at 18 Months
Description: as for outcome 10
Time Frame: Baseline, 18-months (post intervention follow-up)
Population: Participants who completed dietary recalls at all time points (Baseline, 9-weeks, 6-months, and 18 months).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | iSIPsmarter | Patient Education (PE)
Number analyzed (Participants) | 100 | 108
score on a scale | 4.18 [1.45 to 6.92] | 3.21 [0.39 to 6.03]

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the 18-month follow-up data collection
Description: Given the low risk nature of the sugary beverage intervention, adverse events and/or serious adverse events were determined in a non-systematic method, including self-reporting by participants.
Arm/Group | iSIPsmarter | Patient Education (PE)
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/122
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/122
Other Adverse Events (participants affected / at risk) | 0/127 | 0/122

LIMITATIONS AND CAVEATS:
1. The unique rural Appalachian sample and the exclusion of non-English speakers may limit generalizability
2. Females and individuals with 4-year college degrees are over-represented compared to regional census data.
3. Inclusion criteria related to technology acesss and the use of higher-ed recruting partners impact the socio-economic status of the sample
4. Sugar-sweetened beverage intake was self-reported
5. The trial was not powered for secondary outcomes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT05030753/Prot_SAP_000.pdf